CLINICAL TRIAL: NCT05334017
Title: Comparison of the Effect of Xylometazoline and Cocaine on Epistaxis When Administered as Local Vasoconstrictors Prior to Nasal Intubation
Brief Title: Xylometazoline and Cocaine for Nasal Vasoconstriction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mo Haslund Larsen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 89303200; 2021-000691-11 (EudraCT Number); H-21028051 (Other: Regional Committee on Health Research Ethics)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Epistaxis
Keywords: nasal intubation; vasoconstriction; epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylometazoline (Active Comparator): Xylometazoline 0,1% as nasal solution given immediately prior to nasal intubation
  Interventions: Drug: Xylometazoline 0,1%
- Cocaine (Active Comparator): Cocaine 4% as nasal solution given immediately prior to nasal intubation
  Interventions: Drug: Cocaine 4%

INTERVENTIONS:
Drug: Xylometazoline 0,1% — 1 ml of 0,1% xylometazoline diluted with 1 ml of 0,9% isotonic saline solution given as a nasal spray
  Other Names: Zymelin
  Arms: Xylometazoline
Drug: Cocaine 4% — 2 ml of 4% cocaine given as a nasal spray
  Other Names: Cocaine hydrochloride 4%
  Arms: Cocaine

SUMMARY:
The objective of this study is to compare xylometazoline and cocaine's effect on minimizing epistaxis when administered as a local vasoconstrictor prior to nasal intubation.

The investigators hypothesize that there will be a lower bleeding score in the group receiving xylometazoline as compared with the group receiving cocaine.

DETAILED DESCRIPTION:
When performed by trained personnel nasotracheal intubation is a safe and effective technique for attaining a secure airway in preparation for surgery of the head and neck. Upon intubation the nasal mucosa must be sufficiently lubricated and decongested in order to minimize the risk of epistaxis. For this purpose several topical agents are suggested, the most common being adrenaline, cocaine and oxymetazoline/xylometazoline in varying combinations and dosages. As such, no broad consensus or guidelines currently exist on a single recommended drug for the prevention of epistaxis induced by nasal intubation.

In 1990 Katz et. al performed a study comparing three interventions: cocaine, lidocaine with epinephrine and oxymetazoline in regard to the prevention of epistaxis on nasotracheal intubation. This study included 14 patients in each of their three groups and the authors concluded that oxymetazoline and cocaine were equally effective. However, due to their limited sample size that study was clearly inconclusive, and the investigators wish to repeat such a comparison.

The trial drug xylometazoline is commonly used in Danish operating rooms under the registered trademark Zymelin. It is an adrenergic drug typically used for decongestion of the nose and its local vasoconstrictive effect occurs after a few minutes and lasts 10-12 hours. The drug is readily available without prescription and in theory the patient could administer this themselves on their way to surgery. Oxymetazoline used by Katz et. al and xylometazoline used in Danish hospitals have similar decongestive effects as oxymetazoline is a derivative of xylometazoline. The two drugs share pharmacodynamics varying only on receptor subtype affinity in their direct action on alpha-adrenergic receptors in the arterioles of the nasal mucosa. Both drugs result in vasoconstriction that leads to decreased blood flow and thereby decongests the nose.

The second trial drug cocaine is also routinely used. It is a magistral formula used especially due to its unique combination of both vasoconstrictive and analgesic properties. It is a potent vasoconstrictor through its ability to inhibit the reuptake and metabolism of catecholamines, which then in greater concentration produce adrenergic effects. Uniquely cocaine also binds to and blocks axonal membrane sodium channels, thus interfering with the propagation of action potentials and thereby exerting an analgesic effect. When administered in doses thought to avoid systemic effects, cocaine is a safe local anesthetic agent. The recommended dosage varies considerably throughout the literature with safe doses ranging between 1.5-3.0 mg/kg.

The investigators wish to compare the effects of xylometazoline and cocaine regarding their prevention of epistaxis during and immediately after nasal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for nasal intubation
* Proficient in spoken and written Danish

Exclusion Criteria:

* Intubation to be done on awake patient
* Pregnancy

  * Women of childbearing potential must produce a negative hCG urine stix to participate
* Known symptomatic coronary artery disease

  * As declared by patient or noted in the patient's file
* Untreated hypertension

  * As declared by patient or noted in the patient's file
  * Not taking antihypertension drugs
* Hypersensitivity to the active substance or to any of the excipients of Zymelin

  * As declared by patient or noted in the patient's file
* Closed-angle glaucoma

  * As declared by patient or noted in the patient's file

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Bleeding score | Immediately following nasal intubation
  Evaluation of epistaxis measured on a predefined scale of 0-3:
  0. No sign of bleeding
  1. Blood only on the tracheal tube
  2. Pooling of blood in the pharynx
  3. Bleeding to the extent that it complicates intubation

SECONDARY OUTCOMES:
Qualitative measurements of cocaine's main metabolite benzoylecgonine in saliva | Immediately prior to nasal intubation, 60 minutes after administration of cocaine and 24 hours after administration of cocaine.
  For cocaine-group only, saliva samples will be obtained and analyzed on the DrugTest 5000 machine used by the Danish Police Force in order to evaluate pharmacokinetics.
Quantitative measurements of cocaine in whole blood. | Immediately prior to nasal intubation, 60 minutes after administration of cocaine and 24 hours after administration of cocaine.
  In the cocaine group only, blood samples will be drawn and analyzed for the presence of cocaine in order to evaluate pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Mo Haslund Larsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No